CLINICAL TRIAL: NCT02953600
Title: Effect of Cyanobacteria Patients With Chronic Hepatitis B Surface Antigen Quantitative Concentration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N201608026
Record Dates: First submitted 2016-10-27; First posted 2016-11-03 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-10

CONDITIONS: HBV Carrier

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Dose Spirulina Platensis (Experimental): Spirulina platensis pill/500mg, 3 pills before each meal /6 pills per day
  Interventions: Dietary Supplement: Standard Dose Spirulina Platensis
- Zero Spirulina Platensis (Active Comparator): Spirulina platensis pill/500mg, 6 pills before each meal /12 pills per day
  Interventions: Dietary Supplement: Double Dose Spirulina Platensis
- Double Dose Spirulina Platensis (Active Comparator): same as usual, non pill taken
  Interventions: Other: Zero Spirulina Platensis

INTERVENTIONS:
Dietary Supplement: Standard Dose Spirulina Platensis — As previous small scale of clinical trial results in HBV patients provided by Far East Bio-Tec Company, lamivudine combined with oral Spirulina platensis would also improve the sero-conversion rates of HBeAg.
  Arms: Standard Dose Spirulina Platensis
Other: Zero Spirulina Platensis — the zero pill-taken group is a comparison for two other groups.
  Arms: Double Dose Spirulina Platensis
Dietary Supplement: Double Dose Spirulina Platensis — As previous small scale of clinical trial results in HBV patients provided by Far East Bio-Tec Company, lamivudine combined with oral Spirulina platensis would also improve the sero-conversion rates of HBeAg. Hence, the investigators would like to see if the investigators could improve sero-conversion rates much faster by taking double dose of Spirulina platensis.
  Arms: Zero Spirulina Platensis

SUMMARY:
Hepatocellular carcinoma (HCC) is a very severe disease in Taiwan caused 7,000 deaths per year, and majorly about 70% is caused by the chronic hepatitis B virus infection. A repeat, long-term, and severe chronic hepatitis would be more possible progressed into liver cirrhosis and HCC. As previous records, there might be 2% of chronic HBV patient would progress to liver cirrhosis, and 5% of the liver cirrhosis's patients would develop to HCC. In some cases, the HBV patient also might directly develop to HCC without liver cirrhosis phase.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a very severe disease in Taiwan caused 7,000 deaths per year, and majorly about 70% is caused by the chronic hepatitis B virus infection. A repeat, long-term, and severe chronic hepatitis would be more possible progressed into liver cirrhosis and HCC. As previous records, there might be 2% of chronic HBV patient would progress to liver cirrhosis, and 5% of the liver cirrhosis's patients would develop to HCC. In some cases, the HBV patient also might directly develop to HCC without liver cirrhosis phase.

Spirulina platensis is a kind of ancient livings for a 3.5 billions years, and had been recognized as a kind of space food by National Aeronautics and Space Administration(USA) because of containing numerous nutrients, especially vitamin B and beta-carotene. Beta-carotene would convert into vitamin A and help keep health vision, skin, and mucosa. With a rich source of vitamins B, especial B12 which is almost only in meals (animal livers), 1.2 grams of Spirulina platensis daily uptake would be sufficient for a human daily need, and also be a very good source for vegetarians. The investigators add the B12 test in this trial as a secondary endpoint to help monitor the absorption rates of the Spirulina platensis in human. Otherwise, the plant pigments in Spirulina platensis would also have many bioactivities on human healthy. Among these bio-activities of Spirulina platensis would contain anti-virus, anti-cancer, immune modulation, anti-inflammation, anti-oxidant, improve liver abnormality, and liver cirrhosis abilities. As previous small scale of clinical trial results in HBV patients provided by Far East Bio-Tec Company, lamivudine combined with oral Spirulina platensis would also improve the sero-conversion rates of HBeAg.

ELIGIBILITY:
Inclusion Criteria:

* In patients with chronic hepatitis B of taking oral antiviral drugs , and the virus has been detected is less than the amount (HBV DNA <20 IU / ml), aged between 20 years to 75 years .

Exclusion Criteria:

* Patients were allergic to seafood.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
HBsAg(quantitative) | treatment continues for 6 months and checks if HBsAg(quantitative) goes down or remain at the same.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shun Wu, Dr, Study Director — WanFangHospital
Locations (1):
- WanFangH, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No